CLINICAL TRIAL: NCT01844440
Title: Diagnostic of Transient Lower Esophageal Sphincter Relaxation With Combined Impedance and High Resolution Manometry in Patients With GERD.
Acronym: HRM RTSIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CHUBX 2012/25
Record Dates: First submitted 2013-03-01; First posted 2013-05-01 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: Gastroesophageal Reflux Disease
Keywords: GERD; tLESR; impedance; manometry
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- HRM (Experimental)
  Interventions: Procedure: High resolution manometry

INTERVENTIONS:
Procedure: High resolution manometry — Subjects will undergo impedance / manometry recording with solid-state catheter systems, during a 30-min fasting and a 2-hour postprandial periods.

SUMMARY:
The aim of this study is to establish and validate High resolution manometry (HRM) criteria for the definition of transient lower esophageal sphincter relaxations (tLESRs) in gastroesophageal reflux disease (GERD) patients.

DETAILED DESCRIPTION:
tLESRs represent the main mechanism of all types of reflux events. Inhibition of transient lower esophageal sphincter relaxations (tLESRs) has become one of the most relevant therapeutic objectives in patients with reflux symptoms resistant to proton pump inhibitors. HRM is the gold standard for detecting and characterizing tLESR, and could be considered as part of the pharmacological evaluation of new drugs targeting tLESRs. HRM criteria for the objective definition of tLESRs in GERD patients have to be established, as it has been done in healthy patients Subjects will undergo impedance / manometry recording with solid-state catheter systems, during a 30-min fasting and a 2-hour postprandial periods.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 to 75 years old
* GERD documented by :

  * Typical reflux symptoms (heartburn, regurgitations) completely responsive to PPI therapy
  * And/or erosive esophagitis or Barrett's esophagus at endoscopy
  * And/or positive pH 24h monitoring (acid exposure time > 5% or positive symptom association indices)
* Possibility of easily positioned transnasal catheter
* Patients covered by social security
* Subjects must provide written, free and informed consent

Exclusion Criteria:

* Pregnant or lactating women
* History of digestive or thoracic surgery (except appendicectomy)
* Patients unable to stop PPI therapy for 7 days
* Subjects unable to provide written consent, including adult under guardianship and emergency situation
* Simultaneous participation in another study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-04; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
tLESRs characteristics | Inclusion (Day 0)
  To characterize tLESRs defined according following criteria:
  * LES basal pressure (mmHg) defined as LES pressure during relaxation
  * LES minimum pressure during relaxation
  * Duration of the LES relaxation (seconds)
  * Integrated relaxation pressure (4 seconds)
Reflux underlying mechanisms | Inclusion (Day 0)
  To detect every reflux and to determine underlying mechanisms
  * Transient lower esophageal sphincter relaxations (tLESR)
  * Low basal LES pressure (free reflux)
  * Increased abdominal pressure
  * Swallow
  * Another mechanism

CONTACTS AND LOCATIONS:
Overall Officials: Frank ZERBIB, MD-PhD, Principal Investigator — University Hospital, Bordeaux
Locations (3):
- France (3):
  - Service d'hépato-gastroentérologie et oncologie digestive, Bordeaux, Bordeaux
  - Service d'Exploration Fonctionnelle Digestive, Lyon, Lyon
  - Institut des Maladies de l'Appareil Digestif (IMAD), Nantes, Nantes